CLINICAL TRIAL: NCT03217916
Title: Evaluation of Kidney Injury Biomarkers in Women Suffering From Preeclampsia
Brief Title: Kidney Injury Biomarkers in Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Collaborators: Luxor International Hospital (Unknown)
Responsible Party: Principal Investigator, Hisham Ahmed El-Sayed Abou-Taleb, Hisham A. Abou-Taleb, Woman's Health University Hospital, Egypt
Other Study IDs: gemy
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Hypertension, Pregnancy-Induced
Keywords: podocyte glycoprotein; kidney injury; preeclampsia
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia | interventions — Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine sample: 40 ml of a freshly obtained urine specimens will be centrifuged at 1,500 rpm for 10 min within 30 min of collection, aliquoted, and stored at -70°C until assayed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normotensive groups: pregnant women with normal blood pressure
  Interventions: Diagnostic Test: Elisa assay of podocyte glycoprotein in urine
- hypertensive groups: pregnant women with severe preclampsia
  Interventions: Diagnostic Test: Elisa assay of podocyte glycoprotein in urine

INTERVENTIONS:
Diagnostic Test: Elisa assay of podocyte glycoprotein in urine — Biomarkers evaluated in urine specimens including podocyte glycoproteins nephrin and podocalyxin, All biomarkers were measured by ELISA. Assay information for sources of ELISA kits, standard cure range, sample dilution factors, etc.
  All assays will be performed following the manufacture's instructions. All specimens will be measured in duplicate.
  Personnel who performed the assays of analyteswere blinded to the clinical information.

SUMMARY:
we found different pattern of podocyte glycoproteins and kidney injury biomarkers in urine specimens between preeclampsia and pregnancy complicated with chronic hypertention compared with normotensive pregnant controls.abnormally elevayed urine biomarkers in severe preeclampsia were completely or prtially reduced 6-8 weaks after delivery to levels comparable with those of normal pregnant subjects.

DETAILED DESCRIPTION:
Study design:

* Type of the study: Aprospective cross sectional study .All patients will be enrolled in the study after obtaining a written consent.
* Setting: This study will be carried in the Emergency room of Assiut university Hospital &Luxor International Hospital

Statistical Methods:

Inclusion criteria:

* the presence of informed consent
* Prim gravid or multi gravid <5
* age:18-35 ys
* Singleton pregnancy with gestational age >34weeks.

Exclusion criteria:

* Serious maternal illness.
* Smokers
* women with pregnancy complicated by nephritic syndrome, diabetic mellitus, or gestational diabetes
* women known to have renal disease
* oliguria
* Methods :

  200 patients with severe peclampsia will be recorded in Assiut university hospital and luxor international hospital in aperiod of 6 months initial assessement: Blood pressure will be measuerd in ER urine analysis will be done in ER by Urine Dipstick Analysis 40 cases will be randomized selected where urine sample will be collected to analyze the markers to be studied

The women will be subjected to the following:

1. Detailed history taking
2. Clinical examination:

   1. General examination: pulse, temperature, blood pressure, body weight and height, body mass index.
   2. Abdominal examination.
3. obestetric Ultrasonography to calculate gestational age,viability , amniotic fluid ,placental site and to exclude any congenital malformation.
4. Assessemet of renal function :urine output,blood urea,serum creatinine, u/s
5. All routine investigations: C.B.C., Rh, blood grouping, kidney functions tests, liver enzymes.
6. sample collection : Freshly obtained urine specimens were centrifuged at 1,500 rpm for 10 min within 30 min of collection, aliquoted, and stored at _70°C until assayed. Dipstick detection for urine protein, pH, and gravity. Urine protein, pH, gravity, etc. were detected by Dipstick (Uri-Trak-3) in all urine specimens before being aliquoted for storage at _70°C. Urine protein was positive for all study subjects in mild and severe preeclamptic groups.

Biomarkers evaluated in urine specimens including podocyte glycoproteins nephrin and podocalyxin, All biomarkers were measured by ELISA. Assay information for sources of ELISA kits, standard cure range, sample dilution factors, etc.

All assays will be performed following the manufacture's instructions. All specimens will be measured in duplicate.

Personnel who performed the assays of analyteswere blinded to the clinical information.

6. postnatal visits: Postnatal investigation, monitoring and treatment (including after discharge from critical care) Blood pressure

Weekly till the end of puerperium.the postatal visits will iclude:

* Measurement of blood pressure
* U/S kidney
* Askig about urinary symptoms as amout of urine ,colour of urine ,and burning sensation.

Postnatal care will be done according to NICE clinical guidelines at the nearby patients health care centre .the patients will be handed on information sheet containing instructions about postnatal care. the patients will be followed up by telephone to report any abnormalities that may occur

ELIGIBILITY:
Inclusion Criteria:

* the presence of informed consent
* Prim gravid or multi gravid <5
* age:18-35 ys
* Singleton pregnancy with gestational age >34weeks

Exclusion Criteria:

* Serious maternal illness.
* Smokers
* women with pregnancy complicated by nephritic syndrome, diabetic mellitus, or gestational diabetes
* women known to have renal disease
* oliguria

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women attending at the Emergency room of Assiut university Hospital &Luxor International Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Magnitude of renal injury caused by preclampsia | within 6 month postpartum
  the changes in renal chemistry (serum creatinine and blood urea) in pregnant women with severe preclampsia

SECONDARY OUTCOMES:
Apgar score of the deliverd fetus | 1, 5 and 10 minutes after delivery
  standard score to assess fetal status after delivery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Gu Y, Loyd S, Jia X, Groome LJ. Increased urinary levels of podocyte glycoproteins, matrix metallopeptidases, inflammatory cytokines, and kidney injury biomarkers in women with preeclampsia. Am J Physiol Renal Physiol. 2015 Dec 15;309(12):F1009-17. doi: 10.1152/ajprenal.00257.2015. Epub 2015 Oct 14. PMID 26671966
- [Background] Sibai B, Dekker G, Kupferminc M. Pre-eclampsia. Lancet. 2005 Feb 26-Mar 4;365(9461):785-99. doi: 10.1016/S0140-6736(05)17987-2. PMID 15733721
- [Background] Karumanchi SA, Lindheimer MD. Preeclampsia and the kidney: footprints in the urine. Am J Obstet Gynecol. 2007 Apr;196(4):287-8. doi: 10.1016/j.ajog.2007.02.013. No abstract available. PMID 17403396